CLINICAL TRIAL: NCT05721365
Title: The Use and Development of Patient Reported Outcome Measures (PROMs) in the Adoptive Cell Therapy (ACT) Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 22_CPCR_32
Record Dates: First submitted 2023-01-20; First posted 2023-02-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-Infusion: Participants prior to commencing Adoptive Cell Therapy (ACT).
- Acute: Participants either receiving ACT or up to 30 days post treatment.
- Sub-acute: Up to 12 months post ACT.
- Long term follow up: From 12 months post ACT onwards

SUMMARY:
The goals of this observational study is to

1. To develop an Adoptive Cell Therapy (ACT)-specific PROM (Patient Reported Outcome Measure) to assess quality of life and symptomatology
2. To develop guidelines/recommendations for the use of PROMs in ACT trials

Participants will be recruited in four separate stages:

Stage 1: Semi-structured interviews to generate PROM items. Stage 2: Cognitive interviews to ensure that all items are clear and easily understood.

Stage 3: Initial pilot of the draft PROM to enable item reduction and refinement.

Stage 4: Pilot of final PROM to assess acceptability in a clinical setting.

DETAILED DESCRIPTION:
The goals of this observational study is to

1. To develop an Adoptive Cell Therapy (ACT)-specific PROM (Patient Reported Outcome Measure) to assess quality of life and symptomatology
2. To develop guidelines/recommendations for the use of PROMs in ACT trials

Participants will be patients who have taken part in ACT clinical trials.

Stage I - Item generation Approximately 20 participant interviews will be conducted with ACT patients to capture their experiences of receiving ACTs including quality of life, symptom experience, adverse events and other relevant themes that may emerge. The investigators will aim to recruit a minimum of 3 participants in each of the following groups: Pre-infusion; Acute (treatment- 30 days post treatment; Sub-acute- up to 12 months post treatment; Long-term follow-up- from 12 months post treatment onwards. The interviews will be audio recorded and transcribed verbatim. The qualitative data will be analysed thematically and key quotes extracted which will be used to create a draft item list. Interviews will be conducted either in person or virtually depending on national social distancing guidance at the time.

Stage II - Cognitive interviewing Following the creation of a draft item list, approximately 5 participants from Stage I and 3-5 study naïve patients will undergo cognitive interviews to ensure that all items are clear and easily understood. The investigators will also explore patient preferences for the layout of the questionnaire, time recall and overall application issues. Investigators will aim to include a range of participants in each of the four groups outlined above.

Stage III - Item reduction and refinement of the draft ACT-PROM. A draft ACT-PROM, FACT-G and the EORTC PATSATC33 will be administered to approximately 100 participants receiving ACT. Approximately 50 patients will be asked to repeat the draft PROM approximately one week later to assess test-retest reliability. Hierarchical item reduction and Rasch analysis will be used to determine which items should be included in the final ACT-PROM.

Stage IV - Pilot testing The final PROM will be pilot tested with approximately 10 patients to assess its acceptability in the clinic setting. The investigators will aim to include a minimum of two participants in each of the four groups outlined above.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are enrolled on Adoptive Cell Therapy (ACT) trial
2. Aged over 16 (no upper age limit)
3. Ability to understand and communicate in the English language
4. Able to provide written informed consent

Exclusion Criteria:

1. Aged under 16
2. Unable to understand and communicate in the English language
3. Unable to provide written informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer who are enrolled on a Adoptive Cell Therapy (ACT) trial.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Draft Adoptive Cell Therapy Patient Reported Outcome Measure (ACT-PROM) Baseline | 100 participants receiving ACT will complete the PROM upon recruitment,
  Draft PROM pilot tested in stage 3 of the study. Content is determined in the first 2 stages of the study.
Draft Adoptive Cell Therapy Patient Reported Outcome Measure (ACT-PROM) 7 days post baseline | 50 of the 100 participants completing the PROM at baseline will repeat the PROM 1 week later.
  Draft PROM pilot tested in stage 3 of the study. Content is determined in the first 2 stages of the study. This will be compared to baseline to determine test-retest reliability.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-G) | Completed during stage 3 of the study at baseline with the draft PROM.
  Questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Responses are collected using 27 items on a 5 point likert type scale. Total score ranges between 0 and 108 with higher scores indicating higher quality of life. Collected to determine construct validity of the draft PROM.
European Organisation for Research and Treatment of Cancer Satisfaction with Cancer Care Core Questionnaire (EORTC PATSATC33) | Completed during stage 3 of the study at baseline with the draft PROM.
  Satisfaction with cancer care core questionnaire. The questionnaire contains three sections addressing the perceived quality of care provided by doctors, nurses/radiotherapy technicians, and services/care organisation. Responses are collected using 33 items on a 5 point likert type scale. Collected to determine construct validity of the draft PROM.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Thistlethwaite, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No